CLINICAL TRIAL: NCT05560880
Title: The Effects of High Intensity Interval Gait Training vs. Moderate Intensity Continuous Gait Training in Multiple Sclerosis
Brief Title: High Intensity Interval Gait Training in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunter College of City University of New York (Other)
Responsible Party: Principal Investigator, Herbert Karpatkin, Associate professor, Hunter College of City University of New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0261
Record Dates: First submitted 2022-09-22; First posted 2022-09-30 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval gait training (Experimental): subjects will receive 3x/week high intensity interval training for 20 minutes over a 4 week period
  Interventions: Behavioral: High Intensity Interval Gait training
- Moderate intensity continuous gait training (Active Comparator): subjects will receive 3x/week moderate intensity continuous gait training for 20 minutes over a 4 week period
  Interventions: Behavioral: Moderate Intensity Interval gait training

INTERVENTIONS:
Behavioral: High Intensity Interval Gait training — Subjects will walk as fast as they can for 30 seconds, followed by a 60 second seated recovery. They will be guarded by a physical therapist at all times.
  Arms: High Intensity Interval gait training
Behavioral: Moderate Intensity Interval gait training — subjects will walk for 20 minutes at theri best comfortable pace
  Arms: Moderate intensity continuous gait training

SUMMARY:
Over 90% of persons with MS (pwMS) complain of difficulty with walking. High intensity interval gait training (HIIGT), where persons alternate brief periods of walking at high speeds with periods of rest has been found to improve walking in other neurologic diagnoses. However its impact on pwMS is not known. Most gait training in MS is done continuously at a slower pace. The purpose of this study is to compare the effects of HIIGT to traditional Moderate Intensity Continuous Gait Training (MICGT) in pwMS.

DETAILED DESCRIPTION:
Purpose: To determine whether pwMS will have greater improvements in gait with HIIGT as compared to MICGT.

Primary Question: Does HIIGT results in greater improvements in gait parameters in pwMS than MICGT? Secondary question: Will HIIGT result in greater improvements in balance, lower extremity strength, lower extremity range of motion and HR when compared to MICGT in pwMS?

Hypothesis: HIIGT will result in greater improvements in gait parameters in pwMS than MICGT.

Justification: Previous research has shown that MICGT, moderate intensity interval training and high intensity non-gait interval training is effective in pwMS. HIIGT has been shown to be effective in persons with stroke but the effects of HIIGT on pwMS are not known.

Outcomes and dissemination of information: We will present our findings at national conferences and submit manuscripts of our findings to the appropriate peer reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* Persons diagnosed with Multiple Sclerosis.
* The ability to walk for 6 minutes continuously with or without assistive device.
* The ability to read, understand and sign a consent form so that they are able to understand the study we are doing
* Above the age of 18

Exclusion Criteria:

* Any cardiopulmonary, orthopedic, or non-MS neurologic disease as we are only examining the effects of MS and need to rule out the impact of other conditions
* Report of a recent exacerbation. Rationale: the impact of the rationale can interfere with the impact of the independent variables

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Six minute walk test time from before to after the intervention | The test will be administered to all subjects one week before and one week after the intervention.The test will be administered to all subjects one week before and one week after the intervention.
  Subjects will walk for six minutes at their best comfortable pace. They will be guarded by physical therapist for the entire walk. Total distance, distance per minute, and heart rate will be measured.

SECONDARY OUTCOMES:
Change in Functional gait assessment score from before to after the intervention | Will be done in the week before and the week after the intervention.Will be done in the week before and the week after the intervention.
  Used to assess balance during different walking conditions
Change in Hand held dynamometry values from before to after the intervention | Will be done the week before and the week after the intervention.
  Use of the strain gauge to determine lower extremity muscle strength
Change in Multiple sclerosis impact scale 29 from before to afterthe intervention | Performed in the week before and the week after the intervention.
  Quality of life measure where are the subject subjectively rates the impact of multiple sclerosis on their life

CONTACTS AND LOCATIONS:
Locations (1):
- Hunter College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No